CLINICAL TRIAL: NCT02205775
Title: Rosuvastatin for Reduction of Myocardial Damage and Systemic Inflammation During Coronary Angioplasty - The REMEDY Study
Brief Title: Rosuvastatin for Reduction of Myocardial Damage and Systemic Inflammation During Coronary Angioplasty
Acronym: REMEDY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficult recruitment
Sponsor: G. d'Annunzio University (Other)
Collaborators: Working Group Aterosclerosi, Trombosi e Biologia Vascolare (Unknown)
Responsible Party: Principal Investigator, Raffaele De Caterina, Professor, Director - Institute of Cardiology, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-013622-17
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2011-02

CONDITIONS: Stable Coronary Artery Disease Undergoing PCI
MeSH Terms: interventions — Atorvastatin; Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- twice placebo before PCI (Placebo Comparator)
  Interventions: Drug: placebo
- atorvastatin 80 + 40 mg pre PCI (Experimental)
  Interventions: Drug: Atorvastatin
- rosuvastatin 40 + 40 mg before PCI (Experimental)
  Interventions: Drug: Rosuvastatin
- rosuvastatin 5 + ezetimibe 10 mg twice before PCI (Experimental)
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe

INTERVENTIONS:
Drug: Atorvastatin — 80 + 40 mg pre PCI
  Arms: atorvastatin 80 + 40 mg pre PCI
Drug: Rosuvastatin — 40 + 40 mg before PCI
  Arms: rosuvastatin 40 + 40 mg before PCI
Drug: Rosuvastatin — 5 mg twice before PCI (+ 10 mg ezetimibe)
  Arms: rosuvastatin 5 + ezetimibe 10 mg twice before PCI
Drug: Ezetimibe — 10 mg twice before PCI (+ 5 mg rosuvastatin)
  Arms: rosuvastatin 5 + ezetimibe 10 mg twice before PCI
Drug: placebo — twice before PCI
  Arms: twice placebo before PCI

SUMMARY:
Myocardial necrosis is relatively frequent after percutaneous coronary intervention and is associated with higher mortality during the follow-up.

Since anti-inflammatory properties of statins have been demonstrated and the benefit of statins in acute coronary syndromes have been proven, this study aims at testing the hypothesis that the pre-procedural intensive statin treatment reduce the extent of peri-procedural necrosis.

DETAILED DESCRIPTION:
Myocardial necrosis, assessed by creatine kinase-MB (CK-MB) elevation, is relatively frequent after percutaneous coronary intervention (PCI), occurring in up to 40% of cases. Although most patients remain asymptomatic and with no changes in cardiac function, even a mild release of CK-MB is associated with higher mortality during the follow-up. A number of treatment strategies have been proposed to limit myocardial damage during PCI, but procedural ischemic myocardial injury remains the most frequent complication after coronary angioplasty.

Several randomized studies have demonstrated the beneficial effects of therapy with HMG-CoA reductase inhibitors (statins) in patients with already established coronary artery disease or in normal subjects with hypercholesterolemia in primary prevention, and retrospective observational studies have suggested that pre-treatment with statins might reduce the incidence of myocardial infarction after coronary intervention. This benefit was confirmed in patients with non-ST segment elevation acute coronary syndromes (NSTE-ACS) undergoing PCI, who received 80 mg atorvastatin 12 h before PCI, with a further 40-mg pre-procedure, as compared with placebo.

The mechanisms underlying the beneficial effects of statins in ischemic conditions are not completely clear. Previous studies have suggested that the anti-inflammatory effect of statins may play a role, showing that the benefit was higher in patients with high C-reactive protein. Since an inflammatory status before angioplasty, as detected by high levels of C-reactive protein, is associated with a higher risk of peri-procedural myocardial necrosis and adverse cardiac events during the follow-up, the anti-inflammatory effects of statins might contribute to reduce myocardial necrosis, by reducing to the microembolization occurring during coronary intervention. Statin administration also rapidly improves endothelial function. Thus, even short-term treatment with statins (unable to provide LDL reduction persistent enough to decrease the atherosclerotic burden) may have important effects on endothelial function and inflammation. In patients undergoing PCI, reduction of peri-procedural myocardial injury after pre-treatment with statins is paralleled by a concomitant attenuation of post-procedural increase of intercellular cell adhesion molecule-1 (ICAM-1) and E-selectin plasma levels, thus reinforcing the concept that a reduction of endothelial inflammatory response may explain peri-procedural protective effect of statins.

Statins induce heme oxygenase-1 (HO-1) expression in vitro and are reported to have pleiotropic benefits that reduce oxidative stress in the vasculature and in various extravascular tissues Two anti-inflammatory cytokines, interleukin-10 (IL-10) and transforming growth factor-beta, play a critical role in the modulation of immunoinflammatory cell infiltration in the atherosclerotic intima and the mechanism underlying the protective effects of IL-10 against inflammatory cell infiltration involves heme oxygenase-1 (HO-1). Moreover, statins can efficiently increase levels of endothelial progenitor cells (EPCs), contributing to vascular repair, in patients with coronary heart disease and in patients with chronic heart failure, and augment EPC proliferative capacity, in a way similar to vascular endothelial growth factor (VEGF).

Therefore, this study is directed at:

1. documenting whether the immediate pre-procedural administration of a statin at a high dosage may reduce the extent of peri-procedural MI compared with placebo on the background of the best current medical therapy;
2. proving that treatment with rosuvastatin, a hydrophilic statin, at the proposed dosage, is at least comparable (and possibly superior) to atorvastatin at the proposed dosage on top of standard treatment in inducing a significant reduction of peri-procedural damage previously documented with atorvastatin in the presence of a 1-week pre-treatment at 40 mg/day (12);
3. characterizing the relevance of HMG-CoA reductase inhibition (vs largely HMGCoA reductase-independent cholesterol lowering) in this phenomenon;
4. providing a mechanistic explanation for such effects, investigating the role of 1) HO-1 and 2) EPCs in the context of peri-PCI myocardial damage.

ELIGIBILITY:
Inclusion Criteria:

- suspected CAD for which an indication to PCI is given: both patients with stable CAD, and stable post-acute coronary syndromes (ACS), both with ST-segment elevation (STEMI) and without ST-segment elevation (NSTE-ACS) patients, provided that markers of myocardial necrosis (CK-MB, troponins) are stabilized (i.e., with variations <20% in two consecutive measurements obtained at ≥6 h time distance before PCI, according to the universal definition of peri-procedural myocardial infarction).

Exclusion Criteria:

* any previously known increase in liver enzymes (AST, ALT) ascribed to liver dysfunction at baseline;
* history of liver toxicity or myopathy on previous treatment with statins;
* left ventricular ejection fraction <30%;
* renal insufficiency, with creatinine >2 mg/dL at baseline;
* ongoing treatment with high-dose statins (atorvastatin 80 mg/d or rosuvastatin 40 mg/d);
* pregnant or lactating women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
myocardial injury | up to 48 hours
  The proportion of patients with a post-procedural increase of any measured marker of myocardial injury (CK-MB, troponin I or troponin T) above upper normal limits, measured at any of the post-PCI determinations at up to 48 hours

SECONDARY OUTCOMES:
Major adverse cardiac events | 1 month
  The combined occurrence of major adverse cardiac events (MACE), including death, myocardial infarction, stroke or the need for unplanned revascularization from the time of the procedure until the end of a 1-month follow-up.
Serum creatinine | 6, 24 and 48 h
  Any post-procedural increase in serum creatinine or decrease in creatinine clearance (Cockcroft-Gault formula)
HO-1 | 6, 24 and 48 h
  Changes in HO-1 levels/biologic activity among treated groups(only for sites participating in the specific substudies)
endothelial progenitor cells (EPCs) | 6, 24 and 48 h
  Changes in EPC levels/biologic activity among treated groups (only for sites participating in the specific substudies)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele De Caterina, Prof, Principal Investigator — Università G. d'Annunzio
Locations (6):
- Italy (6):
  - SS. Annunziata Hospital, Chieti, CH
  - Fondazione IRCCS Policlinico S. Matteo, Pavia, PV
  - A.O. S. Anna e S. Sebastiano - II Università di Napoli, Caserta
  - Azienda ASL 6 - P. Ospedaliero Livorno, Livorno
  - Ospedale Civile G. Fornaroli, Magenta
  - Azienda Ospedaliera - Ospedale San Paolo, Milan